CLINICAL TRIAL: NCT07338591
Title: Digital vs. Analog Inputs in CAD/CAM Orthodontics: A Comparative Clinical Evaluation of Palatal Expander Fabrication Workflow
Status: Not yet recruiting | Type: Observational
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Other Study IDs: MD.25.06.22
Record Dates: First submitted 2025-12-18; First posted 2026-01-14 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2025-07

CONDITIONS: Transverse Maxillary Deficiency
Keywords: Palatal Expander; Hyrax Expander; CAD/CAM Orthodontics; Digital Workflow; Intraoral Scanning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Fully Analogue Workflow: * Input: Physical impression.
  * Model: Poured in dental stone to produce physical model.
  * Fabrication: Hyrax expander fabricated manually by soldering/brazing components directly on the plaster cast using traditional laboratory techniques.
- Hybrid Workflow: * Input: Physical impression
  * Model: Poured in dental stone to produce physical model.
  * Digitization: Desktop scanning of physical model
  * Fabrication: CAD-designed and 3D-printed appliance (Hyrax-type),
- Fully Digital Workflow: * Input: Intraoral scan (IOS) using an optical scanner
  * Model: Virtual model used directly in design software.
  * Fabrication: CAD-designed and 3D-printed appliance (Hyrax-type),

SUMMARY:
36 patients with unilateral or bilateral cross bite treated with hyrax expanders fabricated through three distinct workflows: fully conventional (physical impression + manual fabrication), hybrid (physical impression + CAD/CAM fabrication), and fully digital (intraoral scanning + CAD/CAM fabrication). To evaluate and compare the clinical fit, workflow efficiency, and patient/clinician satisfaction of palatal expanders fabricated using traditional, hybrid digital, and fully digital workflows.

DETAILED DESCRIPTION:
This randomized, three-arm clinical trial aims to compare the clinical performance and workflow efficiency of tooth-borne palatal expanders fabricated using three different manufacturing workflows: fully conventional, hybrid digital, and fully digital. The study evaluates the impact of these workflows on appliance fit at delivery, efficiency of clinical and laboratory procedures, and patient- and clinician-reported satisfaction.

Following enrollment, participants will be randomly allocated into one of three equal groups using a computer-generated randomization sequence. All appliances used in the study will be Hyrax-type maxillary expanders designed to deliver comparable transverse expansion forces, with differences limited to the fabrication workflow.

In the fully conventional workflow, maxillary impressions will be obtained using conventional impression materials. Dental stone casts will be poured and used directly for appliance fabrication. The Hyrax expander will be manually fabricated on the physical cast using traditional laboratory techniques, including wire bending, band adaptation, and soldering or brazing of the expansion screw and components.

In the hybrid digital workflow, maxillary impressions will also be taken using conventional impression materials and poured in dental stone. The resulting physical casts will then be digitized using a desktop optical scanner. The scanned models will be imported into computer-aided design (CAD) software, where the palatal expander will be digitally designed. Appliance fabrication will be completed using additive manufacturing (3D printing), followed by incorporation of the expansion screw as required.

In the fully digital workflow, maxillary arches will be captured directly using an intraoral optical scanner. The generated virtual models will be used without producing a physical cast. Appliance design will be performed entirely within CAD software, and the Hyrax-type expander will be fabricated using 3D printing technology.

At appliance delivery, clinical evaluation will be performed to assess accuracy of fit, seating on the teeth, need for adjustment, and overall clinical acceptability. Any required chairside modifications will be recorded. Workflow efficiency will be assessed by documenting clinical chairside time, laboratory production time, and the incidence of remakes or significant adjustments.

Patient comfort and acceptance, as well as clinician satisfaction with appliance fit and handling, will be assessed using structured questionnaires. Data collected from all three groups will be compared to determine differences in clinical performance and workflow efficiency among conventional, hybrid, and fully digital fabrication approaches.

ELIGIBILITY:
Inclusion Criteria:

* • Aged between 8 and 13 years with transverse maxillary deficiency ( with unilateral or bilateral crossbite ,with or without anterior cross bite)

  * Indicated for tooth-borne maxillary expansion
  * Good oral hygiene and cooperative behavior
  * No prior orthodontic treatment

Exclusion Criteria:

* • Craniofacial anomalies or syndromes

  * Requirement for surgically assisted expansion
  * Poor oral hygiene or high caries index

Ages: 8 Months to 13 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: A total of 36 participants will be selected from outpatient clinic of orthodontics department (Faculty of Dentistry - Mansoura University). Written consent will be obtained from all legal guardians prior to enrollment.
Sampling Method: Probability Sample
Enrollment: 36 (Estimated)
Dates: Start 2025-12-25 (Estimated); Primary Completion 2027-01-25 (Estimated); Study Completion 2027-07-25 (Estimated)

PRIMARY OUTCOMES:
Clinical Fit and accuracy of expander | Immediately after appliance insertion
  For the clinical fit of the palatal expander at delivery, a 5-point Likert scale could be used by the clinician as follows:
  Score Description
  1. Very poor fit - Significant rocking or instability; requires remake
  2. Poor fit - Major adjustment required (e.g., soldering, bending)
  3. Acceptable fit - Minor chairside adjustments needed
  4. Good fit - Minimal adjustment required
  5. Excellent fit - No adjustment needed, passive and accurate seating

SECONDARY OUTCOMES:
Workflow and Chairside adjustment time | Immediately after appliance insertion
  Time measured in minutes from impression to appliance delivery

OTHER OUTCOMES:
Expansion Efficacy | Through study completion, up to 3 months
  Measurement Method: Transverse dental arch width (mm) at canines / premolars / molars (digital calipers on casts/scans) and Arch length.

CONTACTS AND LOCATIONS:
Locations (1):
- faculty of dentistry , Mansoura university, Al Mansurah, Egypt

IPD SHARING:
Plan to Share IPD: Yes
data with request
Supporting Information: SAP
Time Frame: 3 years
Access Criteria: by request